CLINICAL TRIAL: NCT02255019
Title: MRI in Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: H-2-2010-149
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients will receive a faeces sample kit the first day they meet to MRI. The sample should be taken two days after the MRI scan and sent through the mail. The sample should contain about 5-10 g of faeces and it will be analyzed by ELISA method for calprotectin. Calprotectin is a good marker for the degree of inflammation in the intestines.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD, CD, UC: All patients should either have a known IBD diagnose or suspect of having IBD.

SUMMARY:
The aim of this study is to find an optimal magnetic resonance imaging (MRI) method to examine patients with inflammatory bowel disease (IBD). Patients should furthermore avoid being exposed to unnecessary X-rays and invasive examination.

It is the investigators expectation that this study will benefit to future patients, as they will be offered MRI as the first choice. Hereby, the patients avoid the risks and discomfort associated with x-ray examinations. The aim is that patients with IBD achieve better and earlier treatment and if this is achieved it both benefits patient and public health. An earlier treatment leads to fewer hospitalizations and thereby saving the community money.

The investigators hope is that the investigators study will show that MRI is one of the best tool to examine patients with IBD and that this in future leads MRI to be the first choice in contrary to all examinations with x-ray exposer, unless there is any contraindication to MRI.

DETAILED DESCRIPTION:
IBD is a common term for two chronic diseases, Crohn's disease (CD) and ulcerative colitis (UC). IBD occurs often between the ages of 20-30 years. There are about 25,000 people in Denmark with IBD and diseases incidence and prevalence has increased over the past 20 years [1]. In Denmark, the incidence of CD increased fourfold to 10 per 100,000 inhabitants per years and the incidence of UC doubled to 17 per 100,000 inhabitants per years [2]. Its causes are not completely known but it indicates an interaction between genetic and external factors.

IBD as mentions is a chronic disease which means that it flare up periodically throughout life. Studies show that about 50% at a given time is in clinical remission, 25% had moderate disease activity and 25% have significant disease activity [3]. This means that patients with IBD are more likely to undergo repeatedly examinations to confirm or invalidate disease activity. It is essential for patients that the disease is kept under control so they can maintain a normal working life and a well-functioning social life.

Most studies as when the investigators study began have been in the form of conventional small-bowel follow-through and computed tomographic (CT). A few places in Denmark are beginning to experiment with MRI diagnostics but the method has still no standardized protocol.

There are many advantages by using MRI:

Patients avoid being exposed to X-ray radiation and thus the examination can be carried out repeatedly without any problems. It is especially important for fertile women.

There is no evidence of harmful effects of MRI as opposed to CT scanning, where repeated exposure to X-ray radiation increases the risk of cancer [4].

You could potentially avoid more invasive procedures, thus reducing study duration.

General requested the following highlighted in this project:

Compare the three different MRI scans Compare the clinic with MRI: Calprotectin compared with MRI findings.

The investigators will examine the following hypotheses:

MR enterography can diagnose pathology as well as or better than MRI enteroclysis.

Plain MRI can diagnose pathology as well as or better than MRI enteroclysis. Plain MRI can diagnose pathology as well as or better than MRI enterography.

Method:

This study is carried out as a prospective cross-sectional study (study I-V and a pilot study) in collaboration between radiology department and gastroenterology department at Herlev Hospital. The study recruit both inpatients and outpatients with known or suspected IBD. The main study will include at least 77 patients, while pilot study will include a minimum of 15 patients. Two experienced radiologists in the diagnosis of diseases gastrointestinal will describe the MRI scans. Interpretation of MRI are performed according to a standard table. Studies I-III will be compared to evaluate effectiveness these studies.

Patients will receive a faeces sample kit the first day they meet to MRI. The sample should be taken two days after the MRI scan and sent through the mail. The sample should contain about 5-10 g of faeces and it will be analyzed by ELISA method for calprotectin. Calprotectin is a good marker for the degree of inflammation in the intestines. [5] Analysis of each sample immediately after the reception is too costly. The samples are therefore frozen on the gastroenterology department at Herlev Hospital. When the investigators have collected about 20 samples which is expected to do within one month the samples are analyzed for calprotectin. The material are destroyed immediately after the analysis and can not be used in future research projects.

The study was approved by the Local Committee for Health Research Ethics and the Danish Data Protection Agency.

Study I: Plain MR: Patients undergoing an MRI of the abdomen without oral or IV contrast agent [6]. There are several new studies that show that the diffusion-weighted MRI is good at showing pathology [7-9]. Intravenous buscopan is given in all the studies to reduce peristalsis in the intestines during scan.

Study II: MR enterography: This study is done immediately after study I. Patients from the study I must then take approximately 1.5 l VoLume orally over 1 hour. Previous studies have shown that water alone, taken orally is absorbed very quickly in the intestines and thus does not result in the desired dilation [10-11].

VoLume is an aqueous solution of barium sulfate and it is not reabsorbed by the intestine. The contrast has no immediate side effects, it may in some cases cause constipation. It is crucial for the interpretation of MRI to achieve an optimal dilatation of the intestines. In the end of the scan patients get iv gadolinium. MR enterography is the gold standard in this study.

Study III: MR Enteroclysis (MRE): The above patients will undergo MRE approx. 7 days later. A nasojejunal tube will in placed under fluoroscopy. The radiation that patients are exposed to is minimal and without risk [11-12].

For study II and III should be comparable, it is important that the same amount of fluid is consumed in both studies.

Study IV: This part of the study will consist of a questionnaire-based study of the above patients' experience of the studies II-III [13].

Study V: In this study the calprotectin is compared with study II.

Study VI: Conducted as a pilot study. A small group of patients undergoing an MRI scan with IV contrast, as in substudy II, albeit without prior intake of 1.5 l barium solution. These patients also have an MRI enterografi (which substudy II) 3-7 days later. The results from these two scans are compared.

The study does not include operational or other interventional procedures on the patients involved in the study, and will not be used placebo.

Subjects Minimum 77 subjects in study I-V and minimum 15 subjects in the pilot study are included. All patients should eighter have a known IBD diagnose or suspect IBD. There will not be considered healthy subjects. Participants must be over 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* patients with known or suspected IBD
* age > 18 years

Exclusion Criteria:

* age < 18 years
* low kidney function (eGFR < 30)
* contraindication for MRI (pacemaker, metal in the body, claustrophobia)
* dementia
* severe illness
* pregnancy/lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minimum 77 subjects in study I-V and minimum 15 subjects in the pilot study are included. All patients should eighter have a known IBD diagnose or suspect IBD. There will not be considered healthy subjects. Participants must be over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Inflammation changes in gastrointestinal tract in MRI. | 1 day
  Observe the inflammatory changes in bowel.
evaluate MRI using faecal calprotectin (fC) as a reference standard. | 1-3 days
  MRI is evaluated and fC is received about 3 day after MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Kayalvily J. Nielsen, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Department of Diagnostic Radiology, Herlev, Denmark